CLINICAL TRIAL: NCT06630819
Title: Comparing the Effectiveness of Buccal Infiltration of Different Volumes of Articaine for Extraction of Mandibular Posterior Teeth- A Randomized Clinical Trial.
Brief Title: Buccal Infiltration of Different Volumes of Articaine for Extraction.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Muhammad Atif Saleem Agwan, Assistant Professor, Qassim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 608/45/14624
Record Dates: First submitted 2024-09-24; First posted 2024-10-08 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Buccal Infiltration; Articaine; Anesthesia
Keywords: Buccal infiltration; Articaine
MeSH Terms: interventions — Carticaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Buccal infiltration of 3.6 ml of 4% Articaine
  Interventions: Other: 3.6 ml of 4% Articaine
- Group B (Active Comparator): Buccal infiltration of 1.8 ml of 4% Articaine
  Interventions: Other: 1.8 ml of 4% Articaine

INTERVENTIONS:
Other: 1.8 ml of 4% Articaine — Buccal infiltration of 1.8 ml of 4% Articaine
  Arms: Group B
Other: 3.6 ml of 4% Articaine — Buccal infiltration of 3.6 ml of 4% Articaine.
  Arms: Group A

SUMMARY:
This study compares the effectiveness of two different volumes of buccal infiltration of Articaine for the extraction of mandibular posterior teeth. One group receives buccal infiltration of 1.8 ml of 4% Articaine and the other group receives buccal infiltration of 3.6 ml of 4% Articaine.

DETAILED DESCRIPTION:
The most widely and commonly used injection method for the extraction of mandibular posterior teeth is the inferior alveolar nerve block (IANB) technique. However, various complications like pain during injection, transient facial nerve paralysis, trismus, hematoma, and paresthesia are associated with the inferior alveolar nerve block technique.

Local infiltration technique has been proven as a safer and less painful anesthetic injection technique compared to IANB. Unfortunately, the dense nature of cortical bone in the mandibular posterior region hinders sufficient diffusion of anesthetic solution during infiltration. Thus, to achieve an adequate anesthesia for a painless dental extraction of mandibular posterior teeth by infiltration technique, a strong and effective local anesthetic agent having a deeper penetrating property should be used.

Articaine is one of the most widely used local anesthetic agents. It is more potent and has shown more success rate than Lidocaine and Mepivacaine in providing anesthesia in mandibular and maxillary posterior teeth by buccal infiltration diffusibility.

This study compares the effectiveness of two different volumes of buccal infiltration of Articaine for the extraction of mandibular posterior teeth.

ELIGIBILITY:
Inclusion Criteria:

* All healthy patients (ASA I) or patients with mild systemic disease with no functional limitations (ASA II)
* Patients aged ≥ 18 years of age.
* Patients requiring extraction of mandibular posterior teeth including grossly decayed tooth, grade I mobile tooth, root stumps and indicated for therapeutic reasons.
* Patients not allergic to the drugs or anesthetic agents used in the surgery.

Exclusion Criteria:

* Acute infection at the extraction site.
* Patients indicated for surgical extraction of teeth.
* Patients already taking medications affecting pain assessment.
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-11-24 (Actual); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain | From reflection of mucoperiosteum till delivery of tooth out of socket.
  VAS scale is a validated scale measuring pain with possible score range from 0 (no pain) to 100 (severe pain).
Time of onset of anesthesia | upto 10 minutes
  It will be assessed by probing buccal and lingual soft tissue using a dental explorer every 2 minutes after infiltration using a standard digital stop clock.
Presence or absence of pain | From reflection of mucoperiosteum till delivery of tooth out of socket.
  A 100 mm Numerical rating scale assessing intraoperative pain. Possible score ranges from 0 (no pain) to 100 (worst possible pain).

CONTACTS AND LOCATIONS:
Locations (2):
- Saudi Arabia (2):
  - Qassim University, Buraidah, Al Qassim
  - College of Dentistry, Qassim University, Buraidah

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: Study protocol will be provided only if requested through proper channel with proper justification.